CLINICAL TRIAL: NCT04479852
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study of the Safety and Efficacy of SP-624 in the Treatment of Adults With Major Depressive Disorder
Brief Title: A Study of the Safety and Efficacy of SP-624 in the Treatment of Adults With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sirtsei Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP-624-201
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2024-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SP-624 (Experimental): Daily oral capsule, 20 mg/day
  Interventions: Drug: SP-624
- Placebo (Placebo Comparator): Daily oral capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SP-624 — Oral capsule
  Arms: SP-624
Drug: Placebo — Oral capsule
  Arms: Placebo

SUMMARY:
This is a Phase 2 clinical study evaluating the safety and effectiveness of SP-624 as compared to placebo in the treatment of adults with Major Depressive Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent to participate in the study
* Males and females, aged 18 to 65 years
* In generally good physical health
* Body mass index (BMI) must be between 18 and 40 kg/m2
* Females of reproductive potential and males with partners of reproductive potential must agree to remain abstinent or use adequate and reliable contraception throughout the study and for at least 30 days after the last dose of study drug
* Subjects must meet criteria for moderate to severe Major Depressive Disorder, as confirmed by the Mini International Neuropsychiatric Interview (MINI)
* Willing and able to comply with the study design schedule and other requirements

Exclusion Criteria:

* Female who is pregnant, breastfeeding, or less than six months postpartum at Screening
* History or presence of any clinically significant medical condition, disease, or surgical history that could jeopardize the safety of the subject or validity of the study data, or interfere with the absorption, distribution, metabolism, or excretion of the study drug
* Failure to discontinue all psychoactive medications or psychoactive supplements including antidepressants and mood stabilizers, within a time period prior to Baseline corresponding to at least five half-lives of the medication in question
* Presence of a clinically significant abnormality on physical examination or electrocardiogram (ECG), including a corrected QT interval using Fridericia's formula (QTcF) >450 msec for males and >470 msec for females
* Presence of uncontrolled hypertension, defined as consistent systolic blood pressure (SBP) >160 mmHg or consistent diastolic blood pressure (DBP) >95 mmHg despite present therapy
* Screening laboratory value(s) outside the laboratory reference range that are considered to be clinically significant by the Investigator (clinical chemistry, hematology, coagulation, and urinalysis)
* Screening liver function tests (ALT, AST, Alkaline phosphatase) > 2x the upper limit of normal
* Subjects who, in the opinion of the Investigator, are not suitable candidates for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Rigdon, PhD, Study Director — Sirtsei Pharmaceuticals, Inc.
Locations (39):
- United States (39):
  - Alea Research, Phoenix, Arizona
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - Collaborative Neuroscience Research, Garden Grove, California
  - Pacific Research Partners, Oakland, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Collaborative Neuroscience Research, Torrance, California
  - MCB Clinical Research Centers, Colorado Springs, Colorado
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Innovative Clinical Research, Lauderhill, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Institute for Advanced Medical Research, Alpharetta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - American Medical Research, Chicago, Illinois
  - Capstone Clinical Research, Libertyville, Illinois
  - CBH Health, Gaithersburg, Maryland
  - Midwest Research Group, Saint Charles, Missouri
  - Altea Research Institute, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Hassman Research Institute, Marlton, New Jersey
  - SPRI Clinical Trials, Brooklyn, New York
  - Manhattan Behavioral Medicine, New York, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - Clinical Trials of America, Hickory, North Carolina
  - Midwest Clinical Research Center, Dayton, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigations, Portland, Oregon
  - Oregon Center for Clinical Investigations, Salem, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Donald J. Garcia, Jr., MD, PA, Austin, Texas
  - Future Search Trials of Dallas, Dallas, Texas
  - Red Oak Psychiatry Associates, Houston, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Core Clinical Research, Everett, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SP-624 | Placebo
Started | 163 | 156
Safety Population | 161 | 156
Completed | 133 | 130
Not Completed | 30 | 26

BASELINE CHARACTERISTICS:
Population: Safety population - all subjects who took at least one dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | SP-624 | Placebo | Total
Number analyzed (Participants) | 161 | 156 | 317
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 156 | 154 | 310
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 110 | 211
  Male | 60 | 46 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 21 | 37
  Not Hispanic or Latino | 142 | 135 | 277
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 6 | 10 | 16
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 39 | 32 | 71
  White | 108 | 107 | 215
  More than one race | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 161 | 156 | 317

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 4 in Montgomery Asberg Depression Rating Scale (MADRS) Total Score
Description: The Montgomery Asberg Depression rating scale is a 10-item scale used to assess the severity of depression. Individual items are scored on a 7-point scale (0 to 6). The total score is the sum of individual items, ranging from 0 to 60; where a higher score indicates more depression.
Time Frame: Baseline to Week 4
Population: Modified Intent To Treat population - all subjects who are randomized to receive treatment, receive at least one dose of study drug, and have a Baseline and at least one post-dose efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | SP-624 | Placebo
Number analyzed (Participants) | 132 | 125
Score on a scale | -12.6 (0.83) | -10.8 (0.84)
Statistical Analysis 1: Comparison: SP-624 vs Placebo; Test type: Superiority; p = 0.133, Mixed Models Analysis; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-4.1 to 0.5] — A negative difference favors the SP-624 treatment group, i.e., a greater reduction in MADRS score from baseline

2. Secondary Outcome: Change From Baseline to Week 4 in Clinical Global Impression - Severity (CGI-S) Total Score
Description: The CGI-S is a 7-point scale to rate the severity of the participant's illness at the time of assessment, relative to the clinician's past experience with participants who have the same diagnosis. A score of 1 represents "normal" and 7 represents "most extremely ill".
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | SP-624 | Placebo
Number analyzed (Participants) | 132 | 125
Score on a scale | -1.2 (0.10) | -0.9 (0.10)
Statistical Analysis 1: Comparison: SP-624 vs Placebo; Test type: Superiority; p = 0.059, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to 0.0] — A negative difference favors the SP-624 treatment group, i.e., a greater reduction in CGI-S score from baseline

3. Secondary Outcome: Change From Baseline to Week 4 in the 17-item Hamilton Depression Rating Scale (HAM D-17) Total Score
Description: The 17-item Hamilton Depression rating scale is used to assess the severity of depression. Individual items are scored on either a 3-point (0 to 2) or a 5-point scale (0 to 4), with 0=No difficulty/absent and 4=most severe. The total score is the sum of individual items, ranging from 0 to 52; where a higher score indicates more depression.
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | SP-624 | Placebo
Number analyzed (Participants) | 132 | 125
Score on a scale | -8.3 (0.56) | -7.1 (0.57)
Statistical Analysis 1: Comparison: SP-624 vs Placebo; Test type: Superiority; p = 0.159, Mixed Models Analysis; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.7 to 0.4] — A negative difference favors the SP-624 treatment group, i.e., a greater reduction in HAM-D score from baseline

4. Secondary Outcome: Change From Baseline to Week 4 in the Sheehan Disability Scale (SDS)
Description: The Sheehan Disability Scale is a 3-part scale that measures the degree of disruption on work, social, and family life using an 11-point scale where 0 represents "no disruption" and 10 represents "extreme disruption". Each item (work, social, and family life) can have a score of 0-10. A total global functioning impairment score can be utilized by summing the scores from work, social, and family life scales for a value range from 0 to 30, where a higher score represents a worse outcome, i.e., more disruption on work, social, and family life. In addition to the 11-point scale, participants are asked to indicate the number of days in the past week that were "lost" and numbers of days that were "unproductive". The results of these questions have a range from 0 to 7 and are not included in the overall scale total.
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | SP-624 | Placebo
Number analyzed (Participants) | 131 | 124
Score on a scale | -5.6 (0.52) | -4.6 (0.54)
Statistical Analysis 1: Comparison: SP-624 vs Placebo; Test type: Superiority; p = 0.188, Mixed Models Analysis; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-2.5 to 0.5] — A negative difference favors the SP-624 treatment group, i.e., a greater reduction in SDS score from baseline

5. Secondary Outcome: Change From Baseline to Week 4 in the Quick Inventory of Depressive Symptomology - Self Report (QIDS-SR)
Description: The Quick Inventory of Depressive Symptomology - Self Report (QIDS-SR), is a 16 item self-reported scale where each item has a 4-point scale where 0 represents least impact scores while 3 represents greatest impact scores. Some questions are linked such that the highest score in a group of questions is entered once. For example, there are 4 questions related to sleep and the highest score on any of the 4 sleep items is entered once. The total score ranges from 0 to 27 where a higher score indicates more depression.
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | SP-624 | Placebo
Number analyzed (Participants) | 131 | 124
Score on a scale | -5.0 (0.39) | -4.1 (0.40)
Statistical Analysis 1: Comparison: SP-624 vs Placebo; Test type: Superiority; p = 0.091, Mixed Models Analysis; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-2.0 to 0.2] — A negative difference favors the SP-624 treatment group, i.e., a greater reduction in QIDS score from baseline

6. Secondary Outcome: Change From Baseline to Week 4 in the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF)
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) is a 16 item satisfaction scale where each item has a 5-point scale. A score of 1 represents "very poor satisfaction", while a score of 5 represents "very good satisfaction". Only the first 14 items are summed for a total score that ranges from 14 to 70, where a lower score represents a worse outcome.
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | SP-624 | Placebo
Number analyzed (Participants) | 131 | 124
Score on a scale | 9.5 (1.03) | 7.8 (1.06)
Statistical Analysis 1: Comparison: SP-624 vs Placebo; Test type: Superiority; p = 0.243, Mixed Models Analysis; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [-1.2 to 4.6] — A positive difference favors the SP-624 treatment group, i.e., a greater increase in Q-LES-Q score from baseline

7. Post Hoc Outcome: Female Subjects Change From Baseline Montgomery Asberg Depression Rating Scale Score at Week 4
Description: as for outcome 1
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | SP-624 | Placebo
Number analyzed (Participants) | 84 | 86
Score on a scale | -13.4 (1.05) | -9.4 (1.02)
Statistical Analysis 1: Comparison: SP-624 vs Placebo; Test type: Superiority; p = .008, Mixed Models Analysis; Mean Difference (Final Values) = -3.9, 95% CI 2-sided [-6.8 to -1.0] — A negative difference favors the SP-624 treatment group, i.e., a greater reduction in MADRS score from baseline

8. Post Hoc Outcome: Female Change From Baseline to Week 4 in Clinical Global Impression - Severity (CGI-S) Total Score
Description: as for outcome 2
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | SP-624 | Placebo
Number analyzed (Participants) | 84 | 86
Score on a scale | -1.2 (0.12) | -0.8 (0.11)
Statistical Analysis 1: Comparison: SP-624 vs Placebo; Test type: Superiority; p = 0.006, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.8 to -0.1] — A negative difference favors the SP-624 treatment group, i.e., a greater reduction in CGI-S score from baseline

9. Post Hoc Outcome: Male Subjects Change From Baseline Montgomery Asberg Depression Rating Scale Score at Week 4
Description: as for outcome 1
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | SP-624 | Placebo
Number analyzed (Participants) | 48 | 39
Score on a scale | -11.3 (1.21) | -14.0 (1.35)
Statistical Analysis 1: Comparison: SP-624 vs Placebo; Test type: Superiority; p = 0.134, Mixed Models Analysis; Mean Difference (Final Values) = 2.7, 95% CI 2-sided [-0.8 to 6.3] — A negative difference favors the SP-624 treatment group, i.e., a greater reduction in MADRS score from baseline

10. Post Hoc Outcome: Male Change From Baseline to Week 4 in Clinical Global Impression - Severity (CGI-S) Total Score
Description: as for outcome 2
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | SP-624 | Placebo
Number analyzed (Participants) | 48 | 39
Score on a scale | -1.0 (0.15) | -1.2 (0.16)
Statistical Analysis 1: Comparison: SP-624 vs Placebo; Test type: Superiority; p = 0.437, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.3 to 0.6] — A negative difference favors the SP-624 treatment group, i.e., a greater reduction in CGI-S score from baseline

ADVERSE EVENTS:
Time Frame: Consent through 2 week follow up, up to 10 weeks (up to 28 day screening period, 4 week treatment period, and 2 week follow up period)
Description: Adverse events spontaneously reported by the subject and/or in response to an open question from the study personnel (i.e., how are you feeling?) or revealed by observation were recorded during the study at the investigational site.
Arm/Group | SP-624 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/161 | 0/156
Serious Adverse Events (participants affected / at risk) | 0/161 | 2/156
Other Adverse Events (participants affected / at risk) | 35/161 | 36/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SP-624 (N=161) | Placebo (N=156)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SP-624 (N=161) | Placebo (N=156)
Headache (Nervous system disorders) | 13 (14) | 18 (21)
Nausea (Gastrointestinal disorders) | 9 (9) | 13 (14)
Diarrhea (Gastrointestinal disorders) | 9 (9) | 7 (8)
Anxiety (Psychiatric disorders) | 4 (4) | 1 (2)
Dizziness (Nervous system disorders) | 4 (4) | 9 (9)
Somnolence (Nervous system disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/52/NCT04479852/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/52/NCT04479852/SAP_001.pdf